CLINICAL TRIAL: NCT04722120
Title: Low Contrast Agent and Radiation Dose Protocol Liver CT With Deep-learning-based Contrast Boosting Model in Patients at High Risk for HCC: Prospective, Randomized, Single Blinded - Preliminary Study
Brief Title: Low Contrast Agent and Radiation Dose Protocol for Liver CT in Patients With HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SNUH-2016-2272
Record Dates: First submitted 2016-09-08; First posted 2021-01-25 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: CT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Congresses as Topic; Radiation; Contrast Media

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Participants, investigators, and outcome assessors were all masked to the allocation
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional liver CT (Active Comparator): Underwent conventional liver CT on HCC high-risk patient
  Interventions: Radiation: Conventional CT (radiation); Drug: Conventional CT (contrast agent)
- Double low dose CT (Experimental): Underwent double low dose liver CT with 30% lower radiation dose and 20% contrast media on HCC high-risk patient
  Interventions: Radiation: Low radiation dose CT; Drug: Low contrast dose CT; Other: Deep-learning based contrast boosting algorithms

INTERVENTIONS:
Radiation: Low radiation dose CT — Underwent liver CT with 30% lower radiation dose
  Arms: Double low dose CT
Radiation: Conventional CT (radiation) — Underwent liver CT without change of radiation.
  Arms: Conventional liver CT
Drug: Low contrast dose CT — Underwent liver CT 20% lower dose contrast media.
  Other Names: Low contrast medium dosage
  Arms: Double low dose CT
Drug: Conventional CT (contrast agent) — Underwent liver CT without change of contrast media doses.
  Other Names: Standard contrast medium dosage
  Arms: Conventional liver CT
Other: Deep-learning based contrast boosting algorithms — Applied deep-learning based contrast boosting algorithms on acquired CT images
  Arms: Double low dose CT

SUMMARY:
The purpose of this study is to investigate the image quality and clinical feasibility of double low-dose liver computed tomography using a deep-learning-based iodine contrast boosting algorithm in participants at high risk for hepatocellular carcinoma.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the image quality (CNR, subjective inage quality, vessel and lesion conspicuity) and clinical feasibility (rate of lesion detection) of double low-dose liver computed tomography using a deep-learning-based iodine contrast boosting algorithm in participants at high risk for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Tumor marker (aFP, PIVKA) elevation
* Nodular lesion on USG
* Received RFA for HCC

Exclusion Criteria:

* hypersensitivity at iodine
* GFR under 30
* BMI over 30
* Nursing or pregnant women
* enrolled the other study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Detection rate of solid focal lesion in liver | 12 months after last patient's image work up
  diagnostic performance
Quantitative image quality analysis | Immediate after study enrollement
  Contrast-to-Noise

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No